CLINICAL TRIAL: NCT06700278
Title: Effect of Auricular Acupressure and Peripheral Limb Acupoint Massage on Neuropathic Pain, Activities of Daily Living and Quality of Life in Patients With Spinal Cord Injury
Brief Title: Auricular Acupressure and Limb Massage for Neuropathic Pain in Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202409079RIND
Record Dates: First submitted 2024-11-15; First posted 2024-11-21 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-11

CONDITIONS: Spinal Cord Injury
Keywords: acupressure; neuropathic pain; quality of life; Activities of daily living
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Behavioral: auricular acupressure
- control group (Active Comparator): Routine rehabilitation therapy and body acupoint massage.
  Interventions: Behavioral: body acupoint massage

INTERVENTIONS:
Behavioral: auricular acupressure — auricular acupressure was performed three times daily, with each acupoint massaged for three minutes at an optimal pressure level that induced sensations of soreness, numbness, distension, or mild pain. This was conducted five days a week for three weeks, in addition to regular rehabilitation therapy provided five days per week.The selected auricular acupoints include Shenmen (TF4), Subcortex (AT1), Liver (CO12), and Sympathetic (AH6a).
  Arms: experimental group
Behavioral: body acupoint massage — The control group will receive acupoint massage three times daily, with each acupoint being massaged for three minutes. The applied pressure will be adjusted to induce sensations of soreness, numbness, fullness, or mild pain. The intervention will be conducted five days per week for a total of three weeks. The selected body acupoints include Quchi (LI11), Hegu (LI4), Sanyinjiao (SP6), and Zusanli (ST36).
  Arms: control group

SUMMARY:
This randomized controlled trial included 90 patients with spinal cord injury, divided into an experimental group and a control group (45 each). The experimental group received auricular acupressure alongside rehabilitation therapy, while the control group received body acupoint massage alongside rehabilitation therapy. The intervention targeted specific auricular and body acupoints, performed three times daily, five days a week, for three weeks.

DETAILED DESCRIPTION:
This study is a randomized controlled trial conducted in the rehabilitation ward of National Taiwan University Hospital, using a convenience sampling method. A total of 90 spinal cord injury patients who meet the inclusion criteria will be recruited and randomly assigned to either the experimental group (n=45) or the control group (n=45).

The experimental group will receive auricular acupressure in addition to rehabilitation therapy. The selected auricular acupoints include Shenmen (TF4), Subcortex (AT1), Liver (CO12), and Sympathetic (AH6a).

The control group will receive body acupoint massage in addition to rehabilitation therapy. The selected body acupoints include Quchi (LI11), Hegu (LI4), Sanyinjiao (SP6), and Zusanli (ST36).

Both groups will receive acupoint massage three times daily, with each acupoint being massaged for three minutes. The applied pressure will be adjusted to induce sensations of soreness, numbness, fullness, or mild pain. The intervention will be conducted five days per week for a total of three weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old.
2. Spinal cord injury due to traumatic or non-traumatic reasons.
3. Within one year after spinal cord injury.
4. Spinal cord injuries are classified into ASIA grades B to D.
5. DN4 scale ≥ 4 points and PainDETECT scale ≥ 19 points.
6. Able to communicate in Mandarin and Taiwanese or able to read and write Chinese.

Exclusion Criteria:

1. The auricle and surrounding skin are injured, infected or susceptible.
2. Nerve block surgery has been performed previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Douleur Neuropathique 4 questions(DN4) | Before the intervention and on the 5th, 12th, and 19th days of the intervention.
PainDetect Pain Questionnaire | Before the intervention and on the 5th, 12th, and 19th days of the intervention.

SECONDARY OUTCOMES:
Barthel Index | Before the intervention and on the 5th, 12th, and 19th days of the intervention.
WHOQOL-BREF | Before the intervention and on the 5th, 12th, and 19th days of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Weng YUE CI, Study Chair — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No